CLINICAL TRIAL: NCT01953705
Title: Omega 3 PUFA for the Vascular Component of Age-related Cognitive Decline
Brief Title: n-3 PUFA for Vascular Cognitive Aging
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Gene L. Bowman, ND, MPH, Affiliate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R01AG043398 (NIH); R01AG043398-01A1 (NIH)
Record Dates: First submitted 2013-09-24; First posted 2013-10-01 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Age Related Cognitive Decline; Alzheimer's Disease; Vascular Dementia; Endothelial Dysfunction; Executive Dysfunction
Keywords: omega 3 fatty acids; cognitive decline; MRI; endothelial function; white matter; executive function; prevention; DTI; ASL
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular; Cognitive Dysfunction | interventions — Fish Oils; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omega 3 polyunsaturated fatty acids (Experimental): 1.65 grams of EPA+DHA taken daily over 3 years
  Interventions: Drug: Omega 3 PUFA
- Soybean oil (Placebo Comparator): 1.65 grams of soybean oil taken daily over 3 years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega 3 PUFA — fish oil concentrate standardized to long chain n-3 PUFA content
  Other Names: Fish Oil
  Arms: omega 3 polyunsaturated fatty acids
Drug: Placebo
  Other Names: Soybean Oil
  Arms: Soybean oil

SUMMARY:
Brain scans can help identify changes that appear to increase risk for cognitive decline and dementia. Some of these brain changes are thought to reflect actual damage to the small blood vessels that support normal brain function. This clinical trial will determine whether an omega 3 polyunsaturated fatty acid (PUFA) therapy can promote brain health by supporting the small blood vessels in the brain over 3 years in older adults at high risk for cognitive decline and dementia of Alzheimer's type.

DETAILED DESCRIPTION:
The main objective of this study is to determine if omega 3 PUFA can slow the accumulation of brain MRI derived white matter hyper-intensities (WMH) over 3 years in a population at risk for dementia. This trial is designed to collect preliminary data into the mechanism by which PUFA therapy operates on the brain with special attention to the vascular components.

The randomized, double-blind and controlled trial will rigorously test PUFA effects versus a placebo in non-demented elders over 3 years. This biomarker based trial will enroll 100 elders. Aim 1 will assess PUFA effects on neuroimaging parameter changes. Aim 2 will assess PUFA effects on blood-based biomarkers of endothelial health, and Aim 3 will collect preliminary data on PUFA effects on neuropsychological and functional parameters with special attention to the executive and speed of processing skills and gait speed.

ELIGIBILITY:
Inclusion Criteria:

1. Non-demented or mild cognitive impairment, defined as Clinical Dementia Rating =0 or 0.5 and MMSE >=24.
2. Age 75 and older, male and female
3. Total WMH volume ≥ 5 cc
4. Plasma PUFA index (EPA + DHA) < 110 ug/ml or < 5.5 weight percent
5. Sufficient English language skills to complete all tests
6. Geriatric Depression Scale - 15 < 6 documenting absence of a significant depressive syndrome
7. Sufficient vision and hearing to complete all tests
8. Informant available with frequent (at least 1 hour/day or 1 day/week) contact with subject to verify functional status and CDR rating
9. General health status that will not interfere with the ability to complete the prospective study (these conditions are listed below in the study exclusion list)

Exclusion Criteria:

1. Any dementing illness (AD, vascular dementia, normal pressure hydrocephalus, or Parkinson's disease); dementia defined by CDR ≥ 1, MMSE < 24
2. Significant disease of the CNS such as brain tumor, seizure disorder, subdural hematoma, cranial arteritis
3. Alcohol or substance abuse according to DSM-IV criteria within the last 2 years
4. Major depression, schizophrenia, or other major psychiatric disorder defined by DSM-IV criteria
5. Abnormal labs indicating vitamin B12 deficiency, thyroid disease, or UTI (documented bacterial colonization is acceptable)
6. Unstable or significantly symptomatic CVD (e.g. CAD with frequent angina, CHF with dyspnea at rest)
7. Hypertension: defined as uncontrolled BP > 150/90
8. Clinical symptomatic orthostatic hypotension
9. Diabetes mellitus that requires insulin injections
10. History of cortical stroke
11. Cancer within the last 5 years, with the exception of localized prostate cancer (Gleason Grade < 3) and non-metastatic skin cancers (melanoma).
12. Illness that requires >1 visit /month to a clinician
13. Contraindications to MRI (i.e., heart pacemaker, metal plates or objects in head, , claustrophobia)
14. Medications:

    1. CNS active meds that have not been on stable doses for at least 2 months (cimetidine, beta-blockers, and SSRIs)
    2. Neuroleptics, antiparkinsonian agents, systemic corticosteroids, and narcotic analgesics; in the case where these were used for a self-limited time they must have been discounted for a period of five half-lives prior to baseline visit
    3. Over the counter supplements are not by themselves exclusionary, however, subjects are asked not to change the dosing regimen over the course of the trial unless medically indicated; the presence and dose of these agents are recorded
    4. A baseline screen plasma PUFA > 5.5 weight percent of total fatty acids for EPA+DHA will confirm supplementation of O3PUFA history. If patient indicates regular supplementation with fish oil on phone screen, can wash out for 4 months prior to study visit one.
    5. Cholinesterase inhibitors (i.e., Aricept)
    6. Investigational drugs within five half-lives prior to baseline
    7. Anticoagulation therapy: Vitamin K antagonist: warfarin (Coumadin, jantoven), Factor Xa inhibitors: rivaroxaban (xarelto), fondaparinux (arixtra), dibigatran (pradaxa), apixaban (eliquis); Low molecular weight heparins: dalteparin (fragmin), enoxaparin (lovenox)(Incident use of anticoagulant therapy will exclude further study drug allocation. However, subjects will be asked to complete all follow-up visits.)

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-05; Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
total cerebral white matter hyperintensity volume | annual over 3 years
  quantitative MRI

SECONDARY OUTCOMES:
biomarkers of endothelial health | annual over 3 years
  blood based
total brain atrophy | annual over 3 years
  quantitative MRI
medial temporal lobe atrophy | annual over 3 years
  quantitative MRI
ventricular expansion | annual over 3 years
  quantitative MRI

OTHER OUTCOMES:
trail making test part B | annual over 3 years
  neuropsych
digit symbol WAIS-R | annual over 3 years
  neuropsyh
cerebral blood flow | annual over 3 years
  arterial spin labeling
fractional anisotropy within frontal gyri | annual over 3 years
  diffusion tensor imaging

CONTACTS AND LOCATIONS:
Overall Officials: Gene Bowman, ND, MPH, Principal Investigator — Oregon Health and Science University; Lynne Shinto, ND, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Bowman GL, Dayon L, Kirkland R, Wojcik J, Peyratout G, Severin IC, Henry H, Oikonomidi A, Migliavacca E, Bacher M, Popp J. Blood-brain barrier breakdown, neuroinflammation, and cognitive decline in older adults. Alzheimers Dement. 2018 Dec;14(12):1640-1650. doi: 10.1016/j.jalz.2018.06.2857. Epub 2018 Aug 14. PMID 30120040
- [Background] Alber J, Alladi S, Bae HJ, Barton DA, Beckett LA, Bell JM, Berman SE, Biessels GJ, Black SE, Bos I, Bowman GL, Brai E, Brickman AM, Callahan BL, Corriveau RA, Fossati S, Gottesman RF, Gustafson DR, Hachinski V, Hayden KM, Helman AM, Hughes TM, Isaacs JD, Jefferson AL, Johnson SC, Kapasi A, Kern S, Kwon JC, Kukolja J, Lee A, Lockhart SN, Murray A, Osborn KE, Power MC, Price BR, Rhodius-Meester HFM, Rondeau JA, Rosen AC, Rosene DL, Schneider JA, Scholtzova H, Shaaban CE, Silva NCBS, Snyder HM, Swardfager W, Troen AM, van Veluw SJ, Vemuri P, Wallin A, Wellington C, Wilcock DM, Xie SX, Hainsworth AH. White matter hyperintensities in vascular contributions to cognitive impairment and dementia (VCID): Knowledge gaps and opportunities. Alzheimers Dement (N Y). 2019 Apr 9;5:107-117. doi: 10.1016/j.trci.2019.02.001. eCollection 2019. PMID 31011621
- [Background] Dayon L, Cominetti O, Wojcik J, Galindo AN, Oikonomidi A, Henry H, Migliavacca E, Kussmann M, Bowman GL, Popp J. Proteomes of Paired Human Cerebrospinal Fluid and Plasma: Relation to Blood-Brain Barrier Permeability in Older Adults. J Proteome Res. 2019 Mar 1;18(3):1162-1174. doi: 10.1021/acs.jproteome.8b00809. Epub 2019 Feb 15. PMID 30702894
- [Background] Bowman GL, Dodge HH, Guyonnet S, Zhou N, Donohue J, Bichsel A, Schmitt J, Hooper C, Bartfai T, Andrieu S, Vellas B; MAPT/DSA Study Group. A blood-based nutritional risk index explains cognitive enhancement and decline in the multidomain Alzheimer prevention trial. Alzheimers Dement (N Y). 2019 Dec 28;5:953-963. doi: 10.1016/j.trci.2019.11.004. eCollection 2019. PMID 31921969
- [Background] Hooper C, De Souto Barreto P, Coley N, Causse E, Payoux P, Salabert AS, Cesari M, Andrieu S, Bowman GL, Weiner M, Vellas B. Cross-Sectional Associations of Total Plasma Homocysteine with Cortical beta-Amyloid Independently and as a Function of Omega 3 Polyunsaturated Fatty Acid Status in Older Adults at Risk of Dementia. J Nutr Health Aging. 2017;21(10):1075-1080. doi: 10.1007/s12603-017-0989-x. PMID 29188863
- [Background] Bowman GL, Dodge HH, Mattek N, Barbey AK, Silbert LC, Shinto L, Howieson DB, Kaye JA, Quinn JF. Plasma omega-3 PUFA and white matter mediated executive decline in older adults. Front Aging Neurosci. 2013 Dec 16;5:92. doi: 10.3389/fnagi.2013.00092. eCollection 2013. PMID 24379780
- [Result] Bowman GL, Silbert LC, Dodge HH, Lahna D, Hagen K, Murchison CF, Howieson D, Kaye J, Quinn JF, Shinto L. Randomized Trial of Marine n-3 Polyunsaturated Fatty Acids for the Prevention of Cerebral Small Vessel Disease and Inflammation in Aging (PUFA Trial): Rationale, Design and Baseline Results. Nutrients. 2019 Mar 29;11(4):735. doi: 10.3390/nu11040735. PMID 30934894
- [Derived] Shinto LH, Murchison CF, Silbert LC, Dodge HH, Lahna D, Rooney W, Kaye J, Quinn JF, Bowman GL. omega-3 PUFA for Secondary Prevention of White Matter Lesions and Neuronal Integrity Breakdown in Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2426872. doi: 10.1001/jamanetworkopen.2024.26872. PMID 39088212